CLINICAL TRIAL: NCT05533281
Title: Observation on the Efficacy of Three Antiemetics in Preventing Nausea and Vomiting Caused by Intravenous Tramadol Injection and Postoperative Nausea and Vomiting
Brief Title: Efficacy of Three Antiemetics in Preventing Nausea and Vomiting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Nausea and vomiting
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2022-12

CONDITIONS: Nausea and Vomiting
Keywords: tramadol; nausea and vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Tropisetron; Metoclopramide; Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- tropisetron (Experimental): Troisetron was given 30 minutes in advance, and then tramadol 1.5mg/kg was intravenously injected with a micropump at a constant speed.
  Interventions: Drug: tropisetron
- metoclopramide (Experimental): Metoclopramide was given 30 minutes in advance, and then tramadol 1.5mg/kg was injected intravenously with a micropump at a constant speed.
  Interventions: Drug: metoclopramide
- dexamethasone (Experimental): Dexamethasone was given 30 minutes in advance, and then tramadol 1.5mg/kg was injected intravenously with a micropump at a constant speed.
  Interventions: Drug: dexamethasone
- normal saline (Placebo Comparator): Equal dose of normal saline was given 30 minutes in advance, and then tramadol 1.5mg/kg was given intravenously to ensure constant speed.
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: tropisetron — One tropisetron was given 30 minutes in advance, and then tramadol 1.5mg/kg was intravenously injected with a micropump at a constant speed.
  Arms: tropisetron
Drug: metoclopramide — One dose of metoclopramide was given 30 minutes in advance, and then tramadol 1.5mg/kg was injected intravenously with a micropump at a constant speed.
  Arms: metoclopramide
Drug: dexamethasone — One dose of dexamethasone was given 30 minutes in advance, and then tramadol 1.5mg/kg was injected intravenously with a micropump at a constant speed.
  Arms: dexamethasone
Other: normal saline — Equal dose of normal saline was given 30 minutes in advance, and then tramadol 1.5mg/kg was injected intravenously with a micropump at a constant speed.
  Arms: normal saline

SUMMARY:
To explore the effect of commonly used antiemetic drugs on reducing nausea and vomiting caused by intravenous tramadol injection, so as to reduce the incidence of nausea and vomiting in clinical use of tramadol and provide guidance for the clinical use of tramadol injection

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists classification I-II
* 18.5≤BMI≤28
* Patients who receiving breast and thyroid surgery and requiring general anesthesia and receive PCIA
* Voluntarily and be able to understand and sign the informed consent form

Exclusion Criteria:

* Long-term use of analgesics, psychotropic drugs (including opioids, NSAIDS, antidepressants) history
* History of allergy to opioids
* Patients with a history or family history of epilepsy that has not been controlled by treatment
* Sedatives and antidepressants were used 24 hours before surgery
* Failure to cooperate with the study for any reason or in the opinion of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
NRS score of nausea and vomiting | From before administration to 10min after administration
  NRS score of nausea and vomiting was assessed by numerical rating scale (0-10, 0 representing no nausea and 10 the worst nausea imaginable)

SECONDARY OUTCOMES:
Incidence of postoperative nausea and vomiting | From end of operation to 24 hours after operation
  PONV is recorded according to whether the patient present nausea and vomiting during the follow-up visits after surgery
NRS score of postoperative nausea and vomiting | From end of operation to 24 hours after operation
  NRS score of nausea and vomiting was assessed by numerical rating scale (0-10, 0 representing no nausea and 10 the worst nausea imaginable)
Incidence of extra treatment for postoperative nausea and vomiting | From end of operation to 24 hours after operation
  Incidence of extra treatment for postoperative nausea and vomiting was assessed by whether patient using other treatment for postoperative nausea and vomiting during the the follow-up visits after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Guangyou Duan, MD, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for this study is available from the sponsor on reasonable request through email.
Supporting Information: Study Protocol, SAP, ICF, CSR